CLINICAL TRIAL: NCT05656352
Title: Comparison of Masimo Total Hemoglobin SpHb® Continuous Non-invasive Hemoglobin Monitoring Device With Laboratory Complete Blood Count Measurement Using Venous Sample: A Substudy of the Pregnancy Risk Stratification Innovation and Measurement Alliance Maternal and Newborn Health (PRiSMA MNH) Study
Brief Title: Validation of a Non-invasive Hemoglobin Measurement Device in Pregnancy and Postpartum in Kenya, Pakistan, and Zambia
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Emily Smith, PI, George Washington University
Other Study IDs: SpHb 2022
Record Dates: First submitted 2022-11-02; First posted 2022-12-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Pregnancy, High Risk
Keywords: Hemoglobin; Pregnancy
MeSH Terms: interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Pakistan Cohort
  Interventions: Device: Masimo Total Hemoglobin SpHb® Continuous Non-invasive Hemoglobin Monitoring Device; Diagnostic Test: Complete Blood Count
- Kenya Cohort
  Interventions: Device: Masimo Total Hemoglobin SpHb® Continuous Non-invasive Hemoglobin Monitoring Device; Diagnostic Test: Complete Blood Count
- Zambia Cohort
  Interventions: Device: Masimo Total Hemoglobin SpHb® Continuous Non-invasive Hemoglobin Monitoring Device; Diagnostic Test: Complete Blood Count

INTERVENTIONS:
Device: Masimo Total Hemoglobin SpHb® Continuous Non-invasive Hemoglobin Monitoring Device — Masimo Radical-67® Pulse CO-Oximeter and rainbow® sensors.
Diagnostic Test: Complete Blood Count — The test will be done using venous blood collected in EDTA tubes. Samples will be analyzed within 6 hours of collection or stored at 2 to 8C and analyzed within 24 hours. Analysis will be done using a five-part differential hematology analyzer.

SUMMARY:
Accurate, precise, and comparable hemoglobin measurements is of great importance, both for clinical value in diagnosing anemia and ensuring pregnant women receive appropriate treatment. The Masimo Total Hemoglobin SpHb® is a continuous and non-invasive handheld device with an optical sensor placed on the finger that measures hemoglobin levels using pulse oximetry.

The objective of this study is evaluate the compatibility of hemoglobin measurements between SpHb and the gold standard laboratory-based assessment (complete blood count assessed via five-part autoanalyzer) throughout the course of pregnancy and at six weeks postpartum.

DETAILED DESCRIPTION:
Anemia, a condition that affects an estimated 613 million (33%) women of reproductive age worldwide and is classified as a moderate to severe public health problem in many countries, is a secondary outcome in the PRiSMA MNH study. Three current PRiSMA MNH study sites conduct non-invasive and continuous hemoglobin monitoring with a Masimo device (Kenya, Pakistan, Zambia). Accurate, precise, and comparable hemoglobin measurements is of great importance, both for clinical value in diagnosing anemia and ensuring pregnant women receive appropriate treatment.

The Masimo Total Hemoglobin SpHb® is a continuous and non-invasive handheld device with an optical sensor placed on the finger that measures hemoglobin levels using pulse oximetry. The measurement takes under one minute and does not require blood samples or laboratory testing. These characteristics make it a particularly promising medical technology for low-resource areas.

Previous research studies have found that SpHb is able to accurately detect hemoglobin levels in adult patients with a similar degree of bias and standard deviation to point-of-care (PoC) invasive method (e.g., HemoCue device) measurements. However, high variability in bias and in limits of agreements for the Masimo device was found in a study involving pregnant patients.

The objective of this study is evaluate the compatibility of hemoglobin measurements between SpHb and CBC assessed via 5-part autoanalyzer throughout pregnancy and at six weeks postpartum.

This study is nested in the Pregnancy Risk Stratification Innovation and Measurement Alliance (PRiSMA) Maternal and Newborn Health (MNH) study. PRISMA MNH is a population-based, open-cohort study that seeks to evaluate pregnancy risk factors and their associations with adverse pregnancy outcomes in five countries in sub-Saharan Africa and Southeast Asia. Three study sites (located in Zambia, Kenya, and Pakistan) will participate and collect hemoglobin data at five time points (<20 weeks, 20 weeks, 28 weeks, 36 weeks gestation, and six weeks postpartum). The investigators will measure hemoglobin using a venous blood sample via auto-analyzer (gold standard) and the non-invasive device. The investigators will assess agreement between Masimo total hemoglobin and complete blood count and on a continuous scale using Intraclass Correlation Coefficient and Bland-Altman Analysis. The second objective is to assess agreement between the two measures on a binary scale using Positive Percentage Agreement and Negative Percentage Agreement, Cohen's Kappa, and McNemar Test. On an ordinal scale, agreement will be measured using Weighted Cohen's Kappa and Harrel's Concordance Index. Lastly, the investigators will assess factors that might affect the accuracy of Masimo total hemoglobin using linear mixed models.

ELIGIBILITY:
Inclusion Criteria: Any participant that is eligible for the PRiSMA parent study is also considered eligible for this study. Inclusion criteria for the PRiSMA study is as follows:

1. Lives within the study catchment area;
2. Meets minimum age requirement in study site country:

   * Kenya: 18 years of age or those who meet the criteria of emancipated minors;
   * Pakistan: 15 years of age or those who meet the criteria of emancipated minors;
   * Zambia: 15 years of age;
3. Intrauterine pregnancy <20 weeks gestation verified via ultrasound at enrollment;
4. Provides informed consent.

Exclusion Criteria: Research staff may exclude women from the substudy based on the presence of injury, deformity, tattoo, or birthmark that interferes with Masimo sensor placement or performance or a finger size that does not appropriately fit the device.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant participants from the PRiSMA study
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Hemoglobin (<20 weeks gestation) | <20 weeks gestational age
  Hemoglobin levels will be assessed using the Masimo device and via complete blood count (5 part autoanalyzer) during pregnancy: <20 weeks gestation
Hemoglobin (20 weeks gestation) | 18-25 weeks gestational age
  Hemoglobin levels will be assessed using the Masimo device and via complete blood count (5 part autoanalyzer) during pregnancy: 20 weeks
Hemoglobin (28 weeks gestation) | 26-30 weeks gestational age
  Hemoglobin levels will be assessed using the Masimo device and via complete blood count (5 part autoanalyzer) during pregnancy: 28 weeks
Hemoglobin (36 weeks gestation) | 34 weeks gestational age until delivery
  Hemoglobin levels will be assessed using the Masimo device and via complete blood count (5 part autoanalyzer) during pregnancy: 36 weeks.
Hemoglobin (6 weeks postpartum) | 6-12 weeks postpartum
  Hemoglobin levels will be assessed using the Masimo device and via complete blood count (5 part autoanalyzer) at 6 weeks postpartum

CONTACTS AND LOCATIONS:
Locations (4):
- Kenya Medical Research Institute-Center for Global Health Research, Kisumu, Kenya
- Aga Khan University, Karachi, Pakistan
- Zambia (2):
  - Kamwala District Health Centre, Lusaka
  - Women and Newborn Hospital of the University Teaching Hospitals, Lusaka